CLINICAL TRIAL: NCT02225301
Title: Early Childhood Practitioner's Knowledge and Attitudes Regarding Reporting Child Abuse/Neglect-iLookOut
Brief Title: iLookOut for Child Abuse -Online Learning Module for Early Childcare Providers
Acronym: iLookOut
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin H. Levi, Professor of Humanities & Pediatrics, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-1243; IRB-0376 (Other: Penn State College of medicine)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Child Abuse; Child Neglect; Child Maltreatment
Keywords: Child maltreatment; Child Care; Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iLook Out for Child Abuse (Experimental): The online learning module is an interactive, multi-media, self-paced intervention.
  Interventions: Other: iLook Out for Child Abuse

INTERVENTIONS:
Other: iLook Out for Child Abuse — The online learning module is an interactive, multi-media, self-paced intervention.

SUMMARY:
Phase 1 was a randomized control trial that used a test-retest model to evaluate the impact of iLook Out for Child Abuse, an online, interactive learning module about reporting suspected child abuse. Delivered via a learning management system to early childhood professionals who work with infants and young children, this study assessed iLookOut's effect on 1) knowledge about reporting suspected child abuse; 2) attitudes toward reporting suspected child abuse; and 3) preparedness to protect children at risk.

Findings from Phase 1 were that iLookOut will improved knowledge, changed attitudes, and increase self-reported preparedness of early childhood providers to report suspected child abuse.

Phase 2 of this trial is an open-enrollment study that records pre-/post- data on the same measurements as Phase 1, and is available for use (free of charge) for all childcare providers in Pennsylvania at https://www.ilookoutforchildabuse.com.

DETAILED DESCRIPTION:
Despite their daily interactions with young children, little research has been conducted into early childhood professionals' (ECPs') knowledge of, and attitudes towards, reporting of child abuse/neglect. This study:

1. Evaluates the effectiveness of the online learning module, iLook Out for Child Abuse, created to train and inform early childhood providers about reporting suspected child abuse;
2. Identifies early childhood providers' current knowledge regarding Pennsylvania law on mandated reporting of suspected child abuse;
3. Explores the factors influencing early childhood providers' current knowledge and attitudes;
4. Evaluates the impact of an online educational program on early childhood providers' knowledge, attitudes, and patterns of decision-making regarding mandated reporting of suspected child abuse;
5. To explores the factors influencing the impact of an online educational program on early childhood providers' knowledge and attitudes regarding mandated reporting of suspected child abuse

ELIGIBILITY:
Inclusion Criteria:

* Paid or volunteer staff at childcare facility

Exclusion Criteria:

* Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35000 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge regarding reporting suspected child abuse. | 48 months
  Participants will complete pre- and post-intervention measures regarding reporting suspected child abuse. A sample of Phase 1 participants also repeated knowledge measures 3-6 months post-intervention.

SECONDARY OUTCOMES:
Change in attitudes regarding reporting suspected child abuse. | 48 months
  Participants will complete pre- and post-intervention measures to assess attitudes regarding reporting suspected child abuse. A sample of Phase 1 participants also repeated attitudinal measures 3-6 months post-intervention.

OTHER OUTCOMES:
Evaluation of online learning module. | 48 months
  Participants will complete a post-intervention questionnaire evaluating various aspects of the online learning module. A sample of Phase 1 participants also repeated evaluation measures 3-6 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin H Levi, MD PhD, Principal Investigator — Penn State Milton S. Hershey Medical Center / Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center / Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be available after the study's primary outcomes have been fully analyzed and published.

REFERENCES:
- [Derived] Walsh K, Eggins E, Hine L, Mathews B, Kenny MC, Howard S, Ayling N, Dallaston E, Pink E, Vagenas D. Child protection training for professionals to improve reporting of child abuse and neglect. Cochrane Database Syst Rev. 2022 Jul 5;7(7):CD011775. doi: 10.1002/14651858.CD011775.pub2. PMID 35788913
- [Derived] Yang C, Panlilio C, Verdiglione N, Lehman EB, Hamm RM, Fiene R, Dore S, Bard DE, Grable B, Levi B. Generalizing findings from a randomized controlled trial to a real-world study of the iLookOut, an online education program to improve early childhood care and education providers' knowledge and attitudes about reporting child maltreatment. PLoS One. 2020 Jan 8;15(1):e0227398. doi: 10.1371/journal.pone.0227398. eCollection 2020. PMID 31914147
- [Derived] Mathews B, Yang C, Lehman EB, Mincemoyer C, Verdiglione N, Levi BH. Educating early childhood care and education providers to improve knowledge and attitudes about reporting child maltreatment: A randomized controlled trial. PLoS One. 2017 May 19;12(5):e0177777. doi: 10.1371/journal.pone.0177777. eCollection 2017. PMID 28542285
- See also: Website for iLookOut learning module — https://www.ilookoutforchildabuse.com